CLINICAL TRIAL: NCT00952926
Title: A Prospective Observational Study of Patients With Rectal Cancer After Concomitant Radiation and Chemotherapy
Brief Title: Watchful Waiting. An Observational Study of Patients With Rectal Cancer After Concomitant Radiation and Chemotherapy
Status: Completed | Type: Observational
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: WW
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2019-01

CONDITIONS: Rectal Cancer
Keywords: Watchful Waiting; Rectal cancer; Observation; Avoid operation
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate if operation and permanent stoma can be omitted in patients with cancer in the lower part of the rectum.

DETAILED DESCRIPTION:
Patients entering this study are offered the possibility of avoiding an extensive operation and a permanent stoma.

Over the past 2 years Vejle Hospital examined patients with rectal cancer during their course of treatment and we have developed a method to predict complete response.

Patients in this study are treated with chemotherapy and external irradiation supplemented with an endorectal boost (2 fractions). At the start of treatment and weeks 2, 4, and 6 of the treatment course an endoscopy is performed to evaluate the response. The final evaluation is performed 6 weeks after end of treatment. Patients with complete remission are offered observation. Patients with residual tumor are advised to be operated.

Follow-up is performed every 2 months the first year and every 3 months the second year. 2 follow-up visits are planned for the third year. A yearly follow-up is scheduled for the fourth and fifth year.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically verified adenocarcinoma in the rectum
* Planned APR or ultra low resection
* Primary resectable T2 or T3 tumor
* Distance from anus to lower edge of tumor ≤ 6 cm
* Suited for curative intended radiation and chemotherapy
* Accept taking of biopsy and blood samples for translational research
* Age ≥ 18 years
* Normal function of bone marrow

  * leukocytes ≥ 3 x 10^9/l
  * thrombocytes ≥ 100
* Normal liver function

  * ALAT < 2.5 x upper normal value
  * bilirubin < 2.5 x upper normal value
* Renal function

  * Serum creatinin < 1.5 x upper normal value
* Written and orally informed consent

Exclusion Criteria:

* Other malignant disease within the last 5 years apart from basocellular skin cancer and carcinoma in situ cervicis uteri
* Distant metastases
* Pregnant or breast feeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred from surgical departments in Denmark.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Frequency of local recurrence | 1 year

SECONDARY OUTCOMES:
Frequency of cumulative local recurrence | Up to 5 years
Frequency of distant metastases verified by planned PET/CT scans | Up to 5 years.
Overall survival | Up to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jakobsen, DMSc, Principal Investigator — Vejle Hospital
Locations (1):
- Vejle Hospital, Vejle, Denmark

REFERENCES:
- [Derived] Appelt AL, Ploen J, Harling H, Jensen FS, Jensen LH, Jorgensen JC, Lindebjerg J, Rafaelsen SR, Jakobsen A. High-dose chemoradiotherapy and watchful waiting for distal rectal cancer: a prospective observational study. Lancet Oncol. 2015 Aug;16(8):919-27. doi: 10.1016/S1470-2045(15)00120-5. Epub 2015 Jul 5. PMID 26156652